CLINICAL TRIAL: NCT01393899
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multi-Centre Study To Investigate The Safety And Efficacy Of CP-690,550 For Maintenance Therapy In Subjects With Moderate To Severe Crohn's Disease
Brief Title: The Safety And Efficacy Of Maintenance Therapy With CP-690,550
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3921084; 2011-001754-28 (EudraCT Number)
Record Dates: First submitted 2011-07-12; First posted 2011-07-13 (Estimated); Results first posted 2017-01-09 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2016-11

CONDITIONS: Crohn's Disease
Keywords: tofacitinib; Xeljanz; CP-690,550; maintenance therapy
MeSH Terms: conditions — Crohn Disease | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo BID (Placebo Comparator)
  Interventions: Drug: Placebo
- 5mg BID (Experimental)
  Interventions: Drug: CP-690,550
- 10mg BID (Experimental)
  Interventions: Drug: CP-690,550

INTERVENTIONS:
Drug: Placebo — oral tablets twice daily
  Arms: Placebo BID
Drug: CP-690,550 — oral tablets twice daily
  Arms: 5mg BID
Drug: CP-690,550 — oral tablets twice daily
  Arms: 10mg BID

SUMMARY:
This study investigates safety and efficacy of CP-690,550 in adult patients with moderate to severe Crohn's disease who completed the double-blind induction treatment in Study A3921083 and achieved clinical response-100 and/or clinical remission (CDAI<150) at Week 8.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who met study entry criteria, and who completed Week 8 visit of Induction Study A3921083.
* Subjects who achieve clinical response-100 (reduction in CDAI by 100 points) and/or clinical remission (CDAI<150) in Study A3921083.
* Women of childbearing potential must test negative for pregnancy prior to study enrolment.

Exclusion Criteria:

* Subjects who had major protocol violation (as determined by the Sponsor) in the A3921083 study.
* Subjects likely to require any type of surgery during the study period.
* Fecal culture/toxin assay indicating presence of pathogenic infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (91):
- United States (41):
  - ACMG Endoscopy Center, Anaheim, California
  - ACRI - Phase I, LLC, Anaheim, California
  - Advanced Clinical Research Institute-Phase 1, LLC, Anaheim, California
  - West Coast Clinical Trials, Cypress, California
  - Alliance Clinical Research, Oceanside, California
  - Clinical Research Of The Rockies, Lafayette, Colorado
  - Gasteroenterology Consultants of Clearwater, Clearwater, Florida
  - West Coast Endoscopy Center, Clearwater, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Shands Endoscopy Center, Gainesville, Florida
  - Shands Hospital at the University of Florida, Gainesville, Florida
  - Shands Medical Plaza and Cancer Center, Gainesville, Florida
  - University of Florida - College of Medicine, Gainsville, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Gulfshore Endoscopy Center (Endoscopies Only), Naples, Florida
  - North Florida Gastroenterology Research, LLC, Orange Park, Florida
  - Internal Medicine Specialists, Orlando, Florida
  - Gastroenterology Associates of Central Georgia, LLC, Macon, Georgia
  - Cotton-O'Neil Clinical Research Center, Digestive Health, Topeka, Kansas
  - Chevy Chase Endoscopy Center, Chevy Chase, Maryland
  - Metropolitan Gastroenterology Group, PC, Chevy Chase, Maryland
  - East Ann Arbor Health and Geriatrics Center, Ann Arbor, Michigan
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Center for Digestive Health, Troy, Michigan
  - Surgical Centers of Michigan, Troy, Michigan
  - NYU Langone Nassau Gastroenterology Associates, Great Neck, New York
  - Premier Medical Group of the Hudson Valley, PC, Poughkeepsie, New York
  - Investigational Drug Services - University Hospitals Case Medical Center, Cleveland, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Great Lakes Gastroenterology, Mentor, Ohio
  - Digestive Health Specialists of Tyler, Tyler, Texas
  - Endoscopy Center of Tyler, Tyler, Texas
  - University of Utah HSC, Salt Lake City, Utah
  - Cardiology Consultants, Norfolk, Virginia
  - Digestive & Liver Desease Specialists, Norfolk, Virginia
  - Metropolitan Gastroenterology Group, P C, Washington DC, Virginia
  - The Center for Digestive Health, Milwaukee, Wisconsin
  - Wisconsin Center for Advanced Research - GI Associates, LLC, Milwaukee, Wisconsin
  - Allegiance Research Specialists, Wauwatosa, Wisconsin
  - GI Associates, Wauwatosa, Wisconsin
- Australia (3):
  - Nepean Public Hospital, Kingswood, New South Wales
  - Monash Medical Centre, Clayton, Victoria
  - Royal Melbourne Hospital, Melbourne
- AKH Wien Universitaetsklinik fuer Innere Medizin III, Vienna, Austria
- Bulgaria (2):
  - 4 MBAL Parvo vatreshno otdelenie, Sofia
  - MBAL Sofiamed OOD, Otdelenie po gastroenterologia, Sofia
- Canada (5):
  - Office of Dr. David C. Pearson, Victoria, British Columbia
  - Office of Drs. Ranjith Andrew Singh and Jamie D. Papp,, Victoria, British Columbia
  - PerCuro Clinical Research Ltd., Victoria, British Columbia
  - London Health Sciences Centre - University Hospital, London, Ontario
  - Montreal General Hospital - McGill University Health Centre, Montreal, Quebec
- Czechia (3):
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - Medial Pharma spol.s.r.o. (Pharmacy only), Hradec Králové
  - RDG centrum s.r.o. (Radiology only), Hradec Králové
- France (2):
  - Hopital Huriez CHRU de Lille, Lille
  - Hôpital Haut-Lévêque/Service d hépato-gastroentérologie, Pessac
- Germany (5):
  - Charite - Campus Berlin Mitte, Berlin
  - Charite - Campus Benjamin Franklin, Berlin
  - Charite, Universitaetsmedizin Berlin, Campus Virchow-Klinikum, Berlin
  - Universitaetsklinikum Schleswig-Holstein, Kiel
  - Universitaetsklinikum Ulm, Klinik Fuer Innere Medizin I, Ulm
- General Hospital of Athens "Evangelismos",1st Gastroenterology Department, Kolonaki Athens, Greece
- Hungary (7):
  - Szent Janos Korhaz es Eszak-budai Egyesitett Korhazak/I. Belgyogyaszat es Gastroenterologia, Budapest
  - Pannonia Magánorvosi Centrum Kft, Budapest
  - Laboratorium Kft. Fovarosi és Pest Megyei Mikrobiologiai Laboratorium, Budapest
  - Peterfy Sandor Utcai Korhaz, Rendelointezet es Baleseti Kozpont, I. sz. Belgyogyaszat, Budapest
  - Bugat Pal Korhaz Egeszsegugyi Szolgaltato Kozhasznu Nonprofit Kft.,, Gyöngyös
  - Laboratórium Kft. Somogy Megyei Mikrobiológiai Laboratórium, Kaposvár
  - Clinfan Kft., Szekszárd
- Israel (3):
  - Digestive Disease Institute, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Japan (5):
  - The Hospital of Hyogo College of Medicine, Nishinomiya, Hyōgo
  - National Hospital Organization Sendai Medical Center, Sendai, Miyagi
  - Osaka City University Hospital, Osaka, Osaka
  - Toho University Sakura Medical Center, Chiba
  - Hokkaido P.W.F.A.C Sapporo-Kosei general Hospital, Hokkaido
- Netherlands (2):
  - VU University Medical Center, Amsterdam
  - Academisch Medisch Centrum, Amsterdam
- South Africa (2):
  - Kingsbury Hospital, Cape Town, Western Cape
  - Parklands Medical Centre, Durban
- South Korea (3):
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Division of Gastroenterology, Department of Internal Medicine, Seoul
  - ASAN Medical Center,Division of Gastroenterology,Department of Internal Medicine, Seoul
- Spain (3):
  - Hospital Clinic de Barcelona, Barcelona, Barcelona
  - Comite Etico de Investigacion Clinica, Barcelona
  - Hospital Universitario de La Princesa, Madrid
- Ukraine (3):
  - Donetsk National Medical University n.a M. Gorky, Faculty of Internal Medicine #2, Donetsk
  - Municipal Institution "Odesa Regional Clinical Hospital", Odesa Regional Centre of Gastroenterology., Odesa
  - Medical Clinical Research Center of Medical Center "Health Clinic" LLC, Vinnitsa

REFERENCES:
- [Derived] Panes J, Sandborn WJ, Schreiber S, Sands BE, Vermeire S, D'Haens G, Panaccione R, Higgins PDR, Colombel JF, Feagan BG, Chan G, Moscariello M, Wang W, Niezychowski W, Marren A, Healey P, Maller E. Tofacitinib for induction and maintenance therapy of Crohn's disease: results of two phase IIb randomised placebo-controlled trials. Gut. 2017 Jun;66(6):1049-1059. doi: 10.1136/gutjnl-2016-312735. Epub 2017 Feb 16. PMID 28209624
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921084&StudyName=The%20Safety%20And%20Efficacy%20Of%20Maintenance%20Therapy%20With%20CP-690%2C550%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo (two placebo tablets) to match tofacitinib for oral administration BID for 26 weeks.
- Tofacitinib 5 mg BID: Tofacitinib 5 mg (one placebo tablet and one tofacitinib tablet) for oral administration at a dose of 5 mg BID for 26 weeks.
- Tofacitinib 10 mg BID: Tofacitinib 10 mg (two tofacitinib tablets) for oral administration at a dose of 10 mg BID for 26 weeks.
Period: Overall Study
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Started | 59 | 60 | 61
Completed | 27 | 32 | 38
Not Completed | 32 | 28 | 23
Not completed — Study terminated by sponsor | 1 | 0 | 1
Not completed — Other | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Does not meet entrance criteria | 1 | 0 | 1
Not completed — Lack of Efficacy | 26 | 21 | 16
Not completed — Adverse Event | 1 | 5 | 3

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of all participants who received at least 1 dose of study medication in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID | Total
Number analyzed (Participants) | 59 | 60 | 61 | 180
Age, Customized [Number; unit: Participants]
  Less than or equal to (<=)18 years | 0 | 0 | 0 | 0
  Between 18 and 44 years | 34 | 44 | 40 | 118
  Between 45 and 64 years | 23 | 15 | 20 | 58
  More than or equal to (>=)65 years | 2 | 1 | 1 | 4
Gender [Count of Participants; unit: Participants]
  Female | 32 | 30 | 24 | 86
  Male | 27 | 30 | 37 | 94

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Response-100 (as Defined by a Decrease in Crohn's Disease Activity Index [CDAI] Score of at Least 100 Points From Baseline) or Clinical Remission (CDAI Score Less Than [<]150) at Week 26
Description: Clinical response-100 was defined as a reduction in CDAI score of at least 100 points from baseline of the parent A3921083 study. Clinical remission was a CDAI score <150 points. CDAI is a composite index consisting of a weighted scoring of 8 disease variables: number of liquid or very soft stools, extent of abdominal pain, general well-being, occurrence of extra-intestinal symptoms, need for anti-diarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI score was based partly on entries (7 days before evaluation) from participant's diary kept while on study. CDAI scores range from 0 to approximately 600, higher score indicates higher disease activity.
Time Frame: Week 26
Population: Modified full analysis set (mFAS), defined as all randomized participants who received at least 1 dose of investigational product (ie, active or placebo study medication) in this study and who were randomized into 1 of the tofacitinib (CP-690,550) dose groups in Study A3921083.
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 42 | 43 | 43
Percentage of participants | 38.10 [27.94 to 49.16] | 39.53 [29.39 to 50.46] | 55.81 [44.92 to 66.28]
Statistical Analysis 1: Comparison: Placebo vs Tofacitinib 5 mg BID; Test type: Superiority or Other; Difference in Percentage = 1.44, 80% CI 2-sided [-12.11 to 14.99]
Statistical Analysis 2: Comparison: Placebo vs Tofacitinib 10 mg BID; Test type: Superiority or Other; Difference in Percentage = 17.72, 80% CI 2-sided [4.07 to 31.37]

2. Secondary Outcome: Percentage of Participants With Clinical Response-100 or Clinical Remission at Weeks 4, 8, 12 and 20
Description: Clinical response-100 was defined as a reduction in CDAI score of at least 100 points from baseline of the parent A3921083 study. Clinical remission was a CDAI score <150 points. CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid or very soft stools, extent of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for anti-diarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity.
Time Frame: Weeks 4, 8, 12 and 20
Population: mFAS
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 42 | 43 | 43
Percentage of participants
  Week 4 | 73.81 [63.16 to 82.62] | 74.42 [63.96 to 83.05] | 79.07 [68.98 to 86.96]
  Week 8 | 66.67 [55.69 to 76.37] | 67.44 [56.64 to 76.95] | 58.14 [47.22 to 68.46]
  Week 12 | 50.00 [39.12 to 60.88] | 55.81 [44.92 to 66.28] | 53.49 [42.64 to 64.08]
  Week 20 | 40.48 [30.13 to 51.55] | 39.53 [29.39 to 50.46] | 51.16 [40.38 to 61.86]
Statistical Analysis 1: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 4; Test type: Superiority or Other; Difference in Percentage = 0.61, 80% CI 2-sided [-11.57 to 12.79]
Statistical Analysis 2: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 8; Test type: Superiority or Other; Difference in Percentage = 0.78, 80% CI 2-sided [-12.29 to 13.84]
Statistical Analysis 3: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 12; Test type: Superiority or Other; Difference in Percentage = 5.81, 80% CI 2-sided [-8.04 to 19.67]
Statistical Analysis 4: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 20; Test type: Superiority or Other; Difference in Percentage = -0.94, 80% CI 2-sided [-14.56 to 12.68]
Statistical Analysis 5: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 4; Test type: Superiority or Other; Difference in Percentage = 5.26, 80% CI 2-sided [-6.52 to 17.04]
Statistical Analysis 6: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 8; Test type: Superiority or Other; Difference in Percentage = -8.53, 80% CI 2-sided [-21.94 to 4.88]
Statistical Analysis 7: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 12; Test type: Superiority or Other; Difference in Percentage = 3.49, 80% CI 2-sided [-10.40 to 17.37]
Statistical Analysis 8: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 20; Test type: Superiority or Other; Difference in Percentage = 10.69, 80% CI 2-sided [-3.08 to 24.46]

3. Secondary Outcome: Percentage of Participants Achieving Clinical Response-100 at Weeks 4, 8, 12, 20 and 26
Description: Clinical response-100 was defined as a reduction in CDAI score from baseline of at least 100 points. CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid or very soft stools, extent of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for anti-diarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity.
Time Frame: Weeks 4, 8, 12, 20 and 26
Population: mFAS
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 42 | 43 | 43
Percentage of participants
  Week 4 | 73.81 [63.16 to 82.62] | 72.09 [61.49 to 81.04] | 76.74 [66.45 to 85.02]
  Week 8 | 66.67 [55.69 to 76.37] | 62.79 [51.88 to 72.75] | 58.14 [47.22 to 68.46]
  Week 12 | 50.00 [39.12 to 60.88] | 55.81 [44.92 to 66.28] | 51.16 [40.38 to 61.86]
  Week 20 | 38.10 [27.94 to 49.16] | 39.53 [29.39 to 50.46] | 51.16 [40.38 to 61.86]
  Week 26 | 35.71 [25.77 to 46.74] | 37.21 [27.25 to 48.12] | 55.81 [44.92 to 66.28]
Statistical Analysis 1: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 4; Test type: Superiority or Other; Difference in Percentage = -1.72, 80% CI 2-sided [-14.06 to 10.63]
Statistical Analysis 2: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 8; Test type: Superiority or Other; Difference in Percentage = -3.88, 80% CI 2-sided [-17.15 to 9.40]
Statistical Analysis 3: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 12; Test type: Superiority or Other; Difference in Percentage = 5.81, 80% CI 2-sided [-8.04 to 19.67]
Statistical Analysis 4: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 20; Test type: Superiority or Other; Difference in Percentage = 1.44, 80% CI 2-sided [-12.11 to 14.99]
Statistical Analysis 5: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 26; Test type: Superiority or Other; Difference in Percentage = 1.50, 80% CI 2-sided [-11.88 to 14.87]
Statistical Analysis 6: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 4; Test type: Superiority or Other; Difference in Percentage = 2.93, 80% CI 2-sided [-9.06 to 14.92]
Statistical Analysis 7: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 8; Test type: Superiority or Other; Difference in Percentage = -8.53, 80% CI 2-sided [-21.94 to 4.88]
Statistical Analysis 8: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 12; Test type: Superiority or Other; Difference in Percentage = 1.16, 80% CI 2-sided [-12.74 to 15.06]
Statistical Analysis 9: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 20; Test type: Superiority or Other; Difference in Percentage = 13.07, 80% CI 2-sided [-0.63 to 26.77]
Statistical Analysis 10: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 26; Test type: Superiority or Other; Difference in Percentage = 20.10, 80% CI 2-sided [6.54 to 33.66]

4. Secondary Outcome: Percentage of Participants in Clinical Remission at Weeks 4, 8, 12, 20 and 26
Description: Clinical remission was a CDAI score <150 points. CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid or very soft stools, extent of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for anti-diarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity.
Time Frame: Weeks 4, 8, 12, 20 and 26
Population: mFAS
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 42 | 43 | 43
Percentage of participants
  Week 4 | 52.38 [41.42 to 63.16] | 55.81 [44.92 to 66.28] | 58.14 [47.22 to 68.46]
  Week 8 | 47.62 [36.84 to 58.58] | 48.84 [38.14 to 59.62] | 39.53 [29.39 to 50.46]
  Week 12 | 33.33 [23.63 to 44.31] | 46.51 [35.92 to 57.36] | 34.88 [25.14 to 45.75]
  Week 20 | 30.95 [21.52 to 41.84] | 32.56 [23.05 to 43.36] | 39.53 [29.39 to 50.46]
  Week 26 | 28.57 [19.43 to 39.35] | 37.21 [27.25 to 48.12] | 41.86 [31.54 to 52.78]
Statistical Analysis 1: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 4; Test type: Superiority or Other; Difference in Percentage = 3.43, 80% CI 2-sided [-10.41 to 17.28]
Statistical Analysis 2: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 8; Test type: Superiority or Other; Difference in Percentage = 1.22, 80% CI 2-sided [-12.67 to 15.11]
Statistical Analysis 3: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 12; Test type: Superiority or Other; Difference in Percentage = 13.18, 80% CI 2-sided [-0.31 to 26.67]
Statistical Analysis 4: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 20; Test type: Superiority or Other; Difference in Percentage = 1.61, 80% CI 2-sided [-11.33 to 14.55]
Statistical Analysis 5: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 26; Test type: Superiority or Other; Difference in Percentage = 8.64, 80% CI 2-sided [-4.36 to 21.64]
Statistical Analysis 6: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 4; Test type: Superiority or Other; Difference in Percentage = 5.76, 80% CI 2-sided [-8.04 to 19.56]
Statistical Analysis 7: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 8; Test type: Superiority or Other; Difference in Percentage = -8.08, 80% CI 2-sided [-21.83 to 5.66]
Statistical Analysis 8: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 12; Test type: Superiority or Other; Difference in Percentage = 1.55, 80% CI 2-sided [-11.63 to 14.73]
Statistical Analysis 9: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 20; Test type: Superiority or Other; Difference in Percentage = 8.58, 80% CI 2-sided [-4.64 to 21.81]
Statistical Analysis 10: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 26; Test type: Superiority or Other; Difference in Percentage = 13.29, 80% CI 2-sided [0.15 to 26.43]

5. Secondary Outcome: Percentage of Participants in Clinical Remission at Week 4, 8, 12, 20 and 26 Among Participants in Remission at Baseline of Maintenance Study
Description: as for outcome 4
Time Frame: Weeks 4, 8, 12, 20 and 26
Population: mFAS
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 25 | 28 | 26
Percentage of participants
  Week 4 | 72.00 [57.42 to 83.68] | 78.57 [65.41 to 88.34] | 80.77 [67.23 to 90.34]
  Week 8 | 64.00 [49.20 to 76.97] | 64.29 [50.42 to 76.50] | 50.00 [35.93 to 64.07]
  Week 12 | 40.00 [26.53 to 54.77] | 64.29 [50.42 to 76.50] | 42.31 [28.86 to 56.71]
  Week 20 | 36.00 [23.03 to 50.80] | 42.86 [29.87 to 56.67] | 46.15 [32.36 to 60.43]
  Week 26 | 28.00 [16.32 to 42.58] | 39.29 [26.65 to 53.16] | 50.00 [35.93 to 64.07]
Statistical Analysis 1: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 4; Test type: Superiority or Other; Difference in Percentage = 6.57, 80% CI 2-sided [-8.63 to 21.78]
Statistical Analysis 2: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 8; Test type: Superiority or Other; Difference in Percentage = 0.29, 80% CI 2-sided [-16.63 to 17.20]
Statistical Analysis 3: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 12; Test type: Superiority or Other; Difference in Percentage = 24.29, 80% CI 2-sided [7.19 to 41.38]
Statistical Analysis 4: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 20; Test type: Superiority or Other; Difference in Percentage = 6.86, 80% CI 2-sided [-10.32 to 24.03]
Statistical Analysis 5: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 26; Test type: Superiority or Other; Difference in Percentage = 11.29, 80% CI 2-sided [-5.22 to 27.79]
Statistical Analysis 6: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 4; Test type: Superiority or Other; Difference in Percentage = 8.77, 80% CI 2-sided [-6.41 to 23.95]
Statistical Analysis 7: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 8; Test type: Superiority or Other; Difference in Percentage = -14.00, 80% CI 2-sided [-31.59 to 3.59]
Statistical Analysis 8: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 12; Test type: Superiority or Other; Difference in Percentage = 2.31, 80% CI 2-sided [-15.35 to 19.97]
Statistical Analysis 9: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 20; Test type: Superiority or Other; Difference in Percentage = 10.15, 80% CI 2-sided [-7.41 to 27.71]
Statistical Analysis 10: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 26; Test type: Superiority or Other; Difference in Percentage = 22.00, 80% CI 2-sided [4.96 to 39.04]

6. Secondary Outcome: Percentage of Participants in Sustained Clinical Remission (Defined as Being in Clinical Remission at Both Weeks 20 and 26) in the Maintenance Phase
Description: as for outcome 4
Time Frame: Weeks 20 and 26
Population: mFAS
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 42 | 43 | 43
Percentage of participants | 21.43 [13.37 to 31.71] | 23.26 [14.98 to 33.55] | 39.53 [29.39 to 50.46]
Statistical Analysis 1: Comparison: Placebo vs Tofacitinib 5 mg BID; Test type: Superiority or Other; Difference in Percentage = 1.83, 80% CI 2-sided [-9.75 to 13.40]
Statistical Analysis 2: Comparison: Placebo vs Tofacitinib 10 mg BID; Test type: Superiority or Other; Difference in Percentage = 18.11, 80% CI 2-sided [5.57 to 30.64]

7. Secondary Outcome: Percentage of Participants With Sustained Clinical Response-100 (Defined as Having at Least a Clinical Response-100 at Both Weeks 20 and 26 From the A3921083 Baseline) in the Maintenance Phase
Description: Clinical response-100 was defined as a reduction in CDAI score from baseline of at least 100 points. CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid or very soft stools, extent of abdominal pain, general well-being, occurrence of extra-intestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity.
Time Frame: Weeks 20 and 26
Population: mFAS
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 42 | 43 | 43
Percentage of participants | 33.33 [23.63 to 44.31] | 25.58 [16.95 to 36.04] | 51.16 [40.38 to 61.86]
Statistical Analysis 1: Comparison: Placebo vs Tofacitinib 5 mg BID; Test type: Superiority or Other; Difference in Percentage = -7.75, 80% CI 2-sided [-20.39 to 4.88]
Statistical Analysis 2: Comparison: Placebo vs Tofacitinib 10 mg BID; Test type: Superiority or Other; Difference in Percentage = 17.83, 80% CI 2-sided [4.33 to 31.33]

8. Secondary Outcome: CDAI Score by Week
Description: CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid or very soft stools, extent of abdominal pain, general wellbeing, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity
Time Frame: Baseline and Weeks 4, 8, 12, 20 and 26
Population: mFAS
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 42 | 43 | 43
Score on a scale
  Baseline | 135.05 (69.83) [-112 to 273] | 127.23 (60.46) [-131 to 314] | 133.98 (63.31) [-133 to 198]
  Week 4 | 168.24 (103.18) [-117 to 225] | 133.48 (89.94) [-105 to 241] | 143.45 (84.26) [-132 to 276]
  Week 8 | 171.87 (109.18) [-137 to 474] | 149.78 (99.56) [-126 to 266] | 165.69 (95.46) [-133 to 186]
  Week 12 | 181.38 (108.68) [-152 to 199] | 158.56 (119.41) [-113 to 300] | 152.93 (82.77) [-187 to 148]
  Week 20 | 161.76 (91.65) [-176 to 163] | 151.74 (106.09) [-106 to 164] | 112.32 (85.47) [-203 to 106]
  Week 26 | 137.05 (77.65) | 134.77 (80.22) | 110.77 (76.30)

9. Secondary Outcome: Change From Baseline in CDAI Score by Week
Description: as for outcome 8
Time Frame: Weeks 4, 8, 12, 20 and 26
Population: mFAS
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 42 | 43 | 43
Score on a scale
  Week 4 | 33.17 (76.41) [-112 to 273] | 5.85 (69.52) [-131 to 314] | 11.02 (72.22) [-133 to 198]
  Week 8 | 39.85 (83.68) [-117 to 225] | 20.32 (69.59) [-105 to 241] | 101.96 (101.96) [-132 to 276]
  Week 12 | 52.81 (113.91) [-137 to 474] | 32.29 (88.35) [-126 to 266] | 24.07 (84.46) [-133 to 186]
  Week 20 | 32.44 (96.18) [-152 to 199] | 36.83 (90.92) [-113 to 300] | -14.36 (78.58) [-187 to 148]
  Week 26 | 1.50 (93.91) [-176 to 163] | 17.36 (79.81) [-106 to 164] | -16.35 (75.65) [-203 to 106]
Statistical Analysis 1: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 4; Test type: Superiority or Other; p = 0.0637, Linear mixed-effects model; Adjusted Mean Difference = -30.26, 80% CI 2-sided [-51.10 to -9.42] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 2: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 8; Test type: Superiority or Other; p = 0.3054, Linear mixed-effects model; Adjusted Mean Difference = -21.06, 80% CI 2-sided [-47.43 to 5.31] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 3: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 12; Test type: Superiority or Other; p = 0.1316, Linear mixed-effects model; Adjusted Mean Difference = -42.52, 80% CI 2-sided [-78.57 to -6.48] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 4: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 20; Test type: Superiority or Other; p = 0.5704, Linear mixed-effects model; Adjusted Mean Dofference = -18.01, 80% CI 2-sided [-59.01 to 22.99] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 5: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 26; Test type: Superiority or Other; p = 0.8389, Linear mixed-effects model; Adjusted Mean Difference = -6.00, 80% CI 2-sided [-44.22 to 32.21] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 6: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 4; Test type: Superiority or Other; p = 0.1452, Linear mixed-effects model; Adjusted Mean Difference = -23.56, 80% CI 2-sided [-44.27 to -2.85] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 7: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 8; Test type: Superiority or Other; p = 0.6399, Linear mixed-effects model; Adjusted Mean Difference = -9.61, 80% CI 2-sided [-36.03 to 16.81] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 8: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 12; Test type: Superiority or Other; p = 0.1949, Linear mixed-effects model; Adjusted Mean Difference = -37.00, 80% CI 2-sided [-73.57 to -0.42] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 9: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 20; Test type: Superiority or Other; p = 0.1358, Linear mixed-effects model; Adjusted Mean Difference = -47.74, 80% CI 2-sided [-88.62 to -6.87] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 10: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 26; Test type: Superiority or Other; p = 0.0890, Linear mixed-effects model; Adjusted Mean Difference = -50.38, 80% CI 2-sided [-88.03 to -12.72] — Parameter Type: Adjusted Mean Difference

10. Secondary Outcome: Kaplan-Meier Estimate of the Rate of Time to Relapse
Description: Time to relapse was defined as increase in CDAI of more than (>)100 points from the maintenance phase baseline and a CDAI score of >220 points, or an increase to or above the baseline CDAI score in A3921083. CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid or very soft stools, extent of abdominal pain, general wellbeing, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity.
Time Frame: Weeks 4, 8 12, 20 and 26
Population: mFAS, n=number of participants remaining at risk
Measure: Number (80% Confidence Interval); unit: Percent Probability
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 42 | 43 | 43
Percent Probability
  Week 4 (n=35,38,38) | 14.58 [8.42 to 22.37] | 7.14 [3.15 to 13.34] | 11.63 [6.30 to 18.73]
  Week 8 (n=32,35,32) | 21.90 [14.27 to 30.60] | 14.47 [8.35 to 22.21] | 23.51 [15.73 to 32.21]
  Week 12 (n=24,30,27) | 39.18 [29.40 to 48.80] | 26.69 [18.32 to 35.77] | 31.09 [22.19 to 40.38]
  Week 20 (n=19,22,23) | 51.85 [41.33 to 61.37] | 39.11 [29.35 to 48.74] | 38.95 [29.16 to 48.60]
  Week 26 (n=1,1,2) | 69.59 [48.73 to 83.29] | 50.69 [38.96 to 61.27] | 43.31 [32.60 to 53.54]
Statistical Analysis 1: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 4; Test type: Superiority or Other; Difference in Percentage = -7.44, 80% CI 2-sided [-16.14 to 1.26]
Statistical Analysis 2: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 8; Test type: Superiority or Other; Difference in Percentage = -7.43, 80% CI 2-sided [-18.27 to 3.41]
Statistical Analysis 3: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 12; Test type: Superiority or Other; Difference in Percentage = -12.48, 80% CI 2-sided [-25.68 to 0.72]
Statistical Analysis 4: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 20; Test type: Superiority or Other; Difference in Percentage = -12.73, 80% CI 2-sided [-26.81 to 1.34]
Statistical Analysis 5: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 26; Test type: Superiority or Other; Difference in Percentage = -18.90, 80% CI 2-sided [-39.52 to 1.72]
Statistical Analysis 6: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 4; Test type: Superiority or Other; Difference in Percentage = -2.96, 80% CI 2-sided [-12.39 to 6.48]
Statistical Analysis 7: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 8; Test type: Superiority or Other; Difference in Percentage = 1.61, 80% CI 2-sided [-10.14 to 13.36]
Statistical Analysis 8: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 12; Test type: Superiority or Other; Difference in Percentage = -8.09, 80% CI 2-sided [-21.54 to 5.36]
Statistical Analysis 9: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 20; Test type: Superiority or Other; Difference in Percentage = -12.90, 80% CI 2-sided [-26.99 to 1.19]
Statistical Analysis 10: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 26; Test type: Superiority or Other; Difference in Percentage = -26.28, 80% CI 2-sided [-46.54 to -6.02]

11. Secondary Outcome: Percentage of Participants Achieving a Steroid-Free Clinical Remission at Week 26 of the Maintenance Phase - Among Participants on Steroids at A3921084 Baseline
Description: Clinical remission was a CDAI <150 points. CDAI is a composite index consisting of weighted scoring of 8 disease variables: number of liquid or very soft stools, extent of abdominal pain, general wellbeing, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body eight. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity.
Time Frame: Week 26
Population: mFAS who were on steroids at A3921084 Baseline
Measure: Number (80% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 12 | 11 | 15
Percentage of participants | 16.67 [4.52 to 38.55] | 27.27 [10.48 to 51.08] | 33.33 [17.20 to 53.17]
Statistical Analysis 1: Comparison: Placebo vs Tofacitinib 5 mg BID; Test type: Superiority or Other; Difference in Percentage = 10.61, 80% CI 2-sided [-11.44 to 32.66]
Statistical Analysis 2: Comparison: Placebo vs Tofacitinib 10 mg BID; Test type: Superiority or Other; Difference in Percentage = 16.67, 80% CI 2-sided [-4.15 to 37.49]

12. Secondary Outcome: C-Reactive Protein (CRP) by Week
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline and Weeks 4, 8, 12, 20 and 26
Population: mFAS
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 42 | 43 | 43
milligram per liter (mg/L)
  Baseline | 8.08 (13.88) [-3.3 to 110.6] | 7.08 (10.83) [-37.1 to 63.8] | 8.59 (16.43) [-53.3 to 21.4]
  Week 4 | 16.08 (24.62) [-3.2 to 141.3] | 8.04 (17.36) [-40.3 to 17.5] | 7.62 (15.03) [-14.9 to 26.3]
  Week 8 | 15.80 (28.98) [-4.5 to 74.8] | 8.03 (10.86) [-40.5 to 38.1] | 7.24 (16.48) [-6.7 to 11.4]
  Week 12 | 15.49 (17.80) [-4.6 to 60.0] | 8.19 (11.75) [-34.8 to 43.7] | 5.57 (13.52) [-12.1 to 25.4]
  Week 20 | 15.10 (20.37) [-0.4 to 140.0] | 10.07 (14.56) [-16.6 to 41.3] | 6.52 (18.26) [-11.4 to 8.6]
  Week 26 | 27.70 (41.76) | 13.00 (13.65) | 3.57 (3.55)

13. Secondary Outcome: Change From Baseline in CRP by Week
Description: as for outcome 12
Time Frame: Weeks 4, 8, 12, 20 and 26
Population: mFAS
Measure: Mean (Standard Deviation); unit: milligram per liter (mg/L)
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 42 | 43 | 43
milligram per liter (mg/L)
  Week 4 | 10.66 (19.47) [-3.3 to 110.6] | 0.84 (12.52) [-37.1 to 63.8] | -0.97 (10.81) [-53.3 to 21.4]
  Week 8 | 10.33 (24.33) [-3.2 to 141.3] | 0.96 (9.80) [-40.3 to 17.5] | 1.29 (7.24) [-14.9 to 26.3]
  Week 12 | 11.78 (17.85) [-4.5 to 74.8] | 2.36 (12.15) [-40.5 to 38.1] | 0.39 (3.66) [-6.7 to 11.4]
  Week 20 | 11.48 (19.25) [-4.6 to 60.0] | 2.92 (14.86) [-34.8 to 43.7] | 0.91 (6.75) [-12.1 to 25.4]
  Week 26 | 24.07 (40.90) [-0.4 to 140.0] | 6.62 (13.07) [-16.6 to 41.3] | 0.59 (3.75) [-11.4 to 8.6]
Statistical Analysis 1: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 4; Test type: Superiority or Other; p < 0.0001, Linear mixed-effects model; Adjusted Mean Difference = -0.93, 95% CI 2-sided [-1.34 to -0.53] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 2: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 8; Test type: Superiority or Other; p = 0.0024, Linear mixed-effects model; Adjusted Mean Difference = -0.76, 95% CI 2-sided [-1.24 to -0.28] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 3: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 12; Test type: Superiority or Other; p = 0.0044, Linear mixed-effects model; Adjusted Mean Difference = -0.75, 95% CI 2-sided [-1.26 to -0.24] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 4: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 20; Test type: Superiority or Other; p = 0.0582, Linear mixed-effects model; Adjusted Mean Difference = -0.56, 95% CI 2-sided [-1.13 to 0.02] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 5: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 26; Test type: Superiority or Other; p = 0.0865, Linear mixed-effects model; Adjusted Mean Difference = -0.61, 95% CI 2-sided [-1.31 to 0.09] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 6: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 4; Test type: Superiority or Other; p < 0.0001, Linear mixed-effects model; Adjusted Mean Difference = -0.92, 95% CI 2-sided [-1.32 to -0.52] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 7: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 8; Test type: Superiority or Other; p = 0.0002, Linear mixed-effects model; Adjusted Mean Difference = -0.92, 95% CI 2-sided [-1.40 to -0.45] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 8: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 12; Test type: Superiority or Other; p < 0.0001, Linear mixed-effects model; Adjusted Mean Difference = -1.23, 95% CI 2-sided [-1.75 to -0.71] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 9: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 20; Test type: Superiority or Other; p < 0.0001, Linear mixed-effects model; Adjusted Mean Difference = -1.30, 95% CI 2-sided [-1.87 to -0.74] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 10: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 26; Test type: Superiority or Other; p < 0.0001, Linear mixed-effects model; Adjusted Mean Difference = -1.62, 95% CI 2-sided [-2.30 to -0.95] — Parameter Type: Adjusted Mean Difference

14. Secondary Outcome: Fecal Calprotectin by Week
Description: Fecal calprotectin is an inflammatory marker for the gastrointestinal tract and considered as a measurement of neutrophil migration to the gastrointestinal tract. Higher values indicate more serious inflammation.
Time Frame: Baseline and Weeks 8, 12 and 26
Population: mFAS
Measure: Mean (Standard Deviation); unit: milligrams per kilogram (mg/kg)
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 42 | 43 | 43
milligrams per kilogram (mg/kg)
  Baseline | 380.43 (296.24) [-829.0 to 1416.0] | 351.39 (290.67) [-567.0 to 474.0] | 399.33 (346.98) [-945.0 to 775.0]
  Week 8 | 440.81 (350.71) [-410.0 to 986.0] | 295.39 (272.25) [-517.0 to 523.0] | 283.76 (304.43) [-764.0 to 472.0]
  Week 12 | 441.40 (336.51) [-232.0 to 3426.0] | 351.59 (303.08) [-487.0 to 820.0] | 194.00 (208.50) [-606.8 to 312.28]
  Week 26 | 939.11 (1037.39) | 500.18 (337.83) | 243.76 (219.04)

15. Secondary Outcome: Change From Baseline in Fecal Calprotectin by Week
Description: as for outcome 14
Time Frame: Weeks 8, 12 and 26
Population: mFAS
Measure: Mean (Standard Deviation); unit: milligrams per kilogram (mg/kg)
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 42 | 43 | 43
milligrams per kilogram (mg/kg)
  Week 8 | 69.22 (384.35) [-829.0 to 1416.0] | -59.73 (216.36) [-567.0 to 474.0] | -123.95 (336.67) [-945.0 to 775.0]
  Week 12 | 103.55 (311.15) [-410.0 to 986.0] | -1.81 (228.24) [-517.0 to 523.0] | -107.04 (259.68) [-764.0 to 472.0]
  Week 26 | 579.10 (870.77) [-232.0 to 3426.0] | 154.17 (349.49) [-487.0 to 820.0] | -33.75 (204.25) [-606.8 to 312.28]
Statistical Analysis 1: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 8; Test type: Superiority or Other; p = 0.0566, Linear mixed-effects model; Adjusted Mean Difference = -0.39, 95% CI 2-sided [-0.79 to 0.01] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 2: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 12; Test type: Superiority or Other; p = 0.3144, Linear mixed-effects model; Adjusted Mean Difference = -0.21, 95% CI 2-sided [-0.61 to 0.20] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 3: Comparison: Placebo vs Tofacitinib 5 mg BID; Week 26; Test type: Superiority or Other; p = 0.0434, Linear mixed-effects model; Adjusted Mean Difference = -0.56, 95% CI 2-sided [-1.10 to -0.02] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 4: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 8; Test type: Superiority or Other; p = 0.0050, Linear mixed-effects model; Adjusted Mean Difference = -0.57, 95% CI 2-sided [-0.96 to -0.18] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 5: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 12; Test type: Superiority or Other; p = 0.0017, Linear mixed-effects model; Adjusted Mean Difference = -0.66, 95% CI 2-sided [-1.06 to -0.25] — Parameter Type: Adjusted Mean Difference
Statistical Analysis 6: Comparison: Placebo vs Tofacitinib 10 mg BID; Week 26; Test type: Superiority or Other; p < 0.0001, Linear mixed-effects model; Adjusted Mean Difference = -1.20, 95% CI 2-sided [-1.72 to -0.67] — Parameter Type: Adjusted Mean Difference

16. Secondary Outcome: Tofacitinib Plasma Concentration by Nominal Post-Dose Sampling Time and Tofacitinib Dose
Description: Plasma samples were collected from participants for the determination of tofacitinib concentrations. Only samples from tofacitinib-treated participants were subsequently analyzed. Plasma concentration data are summarized by nominal sample collection times specified in the protocol, and actual sample collection times may be different.
Time Frame: Pre-dose, 20 minutes, 40 minutes, 1 hour and 2 hours post-dose at Weeks 12 and 26/early termination visit
Population: Pharmacokinetic analysis set - included all participants who received at least 1 dose of study medication and had at least 1 measurable plasma concentration. n=number of observations above lower limit of quantification.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Number analyzed (Participants) | 48 | 48
nanograms per milliliter (ng/mL)
  Week 12, 0 hours (n=43, 40) | 6.059 (7.4264) [0.000 to 28.7] | 6.832 (5.7271) [0.000 to 20.5]
  Week 12, 20 minutes (n=45, 40) | 31.56 (21.904) [0.120 to 76.4] | 58.53 (53.579) [0.000 to 156]
  Week 12, 40 minutes (n=47, 41) | 47.05 (23.904) [0.685 to 96.1] | 85.23 (43.726) [1.53 to 155]
  Week 12, 1 hour (n=46, 42) | 46.84 (20.365) [6.15 to 95.9] | 82.08 (33.779) [6.12 to 158]
  Week 12, 2 hour (n=44, 42) | 36.52 (14.810) [1.38 to 83.1] | 69.79 (23.274) [24.0 to 134]
  Week 26/ET, 0 hours (n=43, 46) | 6.183 (13.673) [0.000 to 87.5] | 9.510 (17.115) [0.000 to 113]
  Week 26/ET, 20 minutes (n=45, 48) | 40.98 (31.713) [0.000 to 117] | 60.48 (51.084) [0.218 to 167]
  Week 26/ET, 40 minutes (n=46, 48) | 55.83 (44.421) [0.000 to 285] | 85.66 (37.983) [9.87 to 196]
  Week 26/ET, 1 hour (n=45, 48) | 52.59 (42.291) [0.000 to 293] | 86.25 (30.948) [11.4 to 187]
  Week 26/ET, 2 hours (n=44, 48) | 39.09 (22.606) [0.000 to 143] | 64.15 (23.499) [21.9 to 150]

ADVERSE EVENTS:
Time Frame: SAEs were assessed from informed consent through and including 28 calendar days after last administration of study treatment (30 weeks). Non-SAEs were recorded from time of first dose of study treatment through last participant visit (30 weeks).
Description: The same event may appear as both an adverse event (AE) and an SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | Tofacitinib 5 mg BID | Tofacitinib 10 mg BID
Serious Adverse Events (participants affected / at risk) | 7/59 | 6/60 | 8/61
Other Adverse Events (participants affected / at risk) | 28/59 | 40/60 | 35/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=59) | Tofacitinib 5 mg BID (N=60) | Tofacitinib 10 mg BID (N=61)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 3 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal fistula (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Abortion induced (Surgical and medical procedures) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=59) | Tofacitinib 5 mg BID (N=60) | Tofacitinib 10 mg BID (N=61)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 5
Abdominal pain (Gastrointestinal disorders) | 2 | 5 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 2 | 0
Crohn's disease (Gastrointestinal disorders) | 10 | 11 | 7
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 5
Dyspepsia (Gastrointestinal disorders) | 3 | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 2
Toothache (Gastrointestinal disorders) | 0 | 0 | 2
Asthenia (General disorders) | 0 | 2 | 0
Chest pain (General disorders) | 0 | 0 | 2
Fatigue (General disorders) | 1 | 2 | 1
Pyrexia (General disorders) | 2 | 2 | 4
Bronchitis (Infections and infestations) | 0 | 3 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 3
Folliculitis (Infections and infestations) | 0 | 0 | 3
Gastroenteritis (Infections and infestations) | 0 | 2 | 3
Herpes zoster (Infections and infestations) | 0 | 0 | 2
Influenza (Infections and infestations) | 2 | 5 | 3
Nasopharyngitis (Infections and infestations) | 4 | 11 | 5
Oral herpes (Infections and infestations) | 2 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 1
Tooth abscess (Infections and infestations) | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1
Urinary tract infection (Infections and infestations) | 4 | 6 | 8
Vaginal infection (Infections and infestations) | 0/32 | 0/30 | 1/24
Vulvovaginal mycotic infection (Infections and infestations) | 0/32 | 0/30 | 1/24
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 0
Blood creatinine increased (Investigations) | 0 | 2 | 0
Blood pressure increased (Investigations) | 0 | 0 | 2
Lymphocyte count decreased (Investigations) | 0 | 2 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 6 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Headache (Nervous system disorders) | 2 | 4 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 2
Endometriosis (Reproductive system and breast disorders) | 0/32 | 0/30 | 1/24
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less